CLINICAL TRIAL: NCT02662270
Title: Quantitative and Qualitative EEG From Fibromyalgia Patients for the Identification of Abnormal Patterns on Closed Eyes EEG
Brief Title: QEEG and Qualitative EEG for the Identidification of Abnormal Patterns in Fibromyalgia Patients
Acronym: QEEGFP
Status: Completed | Type: Observational
Sponsor: Spanish Foundation for Neurometrics Development (Other)
Collaborators: Universidad de Murcia (Other)
Responsible Party: Sponsor
Other Study IDs: Fibromyalgia and TDCs
Record Dates: First submitted 2016-01-19; First posted 2016-01-25 (Estimated); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; QEEG; Brain activity; fMRI; Diagnosis
MeSH Terms: conditions — Fibromyalgia; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cases: Patients with a fibromyalgia diagnosis established according to the American College of Rheumatology current criteria by a trained physician.
- Controls: Healthy subjects paired by age and gender to the subjects in the cases group.

SUMMARY:
Fibromyalgia is a relatively young condition recently recognized by the WHO as a separated clinical entity. Part of the medical comunity thinks of it as a mixed condition between depresion and rheumatic pain, however, functional data provided by sophisticated imaging techniques points at a diminished brain activity in several brain regions. The present study aims to characterize those findings by means of QEEG in order to establish the electroencephalographic characteristics of fibromyalgia patients.

DETAILED DESCRIPTION:
Fibromyalgia is a disease that part of the general population and even the medical community views with skepticism and only recently was accepted as a true condition by the World Health Organization. Some physicians see it as a form of depresion mixed with rheumatic pain. However recent findings in functional magnetic resonance imaging and positron emited tomography documented diminished brain activity on several regions. The impairments must be located within the areas with a documented functional defect, wherein, spontaneous braincells activity chould arise. Therefor electroencephalography findings should be a valuable diagnostic tool for early detection in fibromyalgia. The present study aims to analyse the differences between bioelectric characteristics in EEG from fibromyalgia patients with their eyes closed in a 21 electrode arragement. Normal graphoelements as well as abnormal ones and its topographic distribution and functional conections will be analyzed.

The working hypotesis is that fibromyalgia patients will present distintive characteristics in the same areas where a diminished brain activity has been documented by metabolic and morphologic tests as a group and that those characteristics are suitable to be measured by QEEG and distinguishable from healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 20 and 70 years old, diagnosed with fibromyalgia and a control group matched by age and gender

Exclusion Criteria:

* Any other concomitant neurologic disease or impairment

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and women between 20 and 70 years old divided in two groups, one consisting in 50 subjects diagnosed with fibromyalgia acording to the current criteria of the American College of Rheumatology and a control group matched by age and gender without fibromyalgia
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-03-12 (Actual)

PRIMARY OUTCOMES:
Differences between groups in Fast Fourier Transformation | Up to one year
  Changes in Power in EEG over different electrodes
Topographic distribution of the frequency bands | Up to one year
  Brain areas with a characteristic pattern
Dominant EEG frequency localization | Up to one year
  To document the dominant frequency in the resting EEG for all subjects
Abnormal EEG-graphoelements description | Up to one year
  To identify the abnormal EEG-graphoelements found in fibromyalgia patients
Functional conectivity | Up to one year
  To identify the different brain connections between fibromyalgia patients

CONTACTS AND LOCATIONS:
Overall Officials: Moises Aguilar-Domingo, PhD, Principal Investigator — Brainmech Foundation
Locations (1):
- Universidad de Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Branco J, Atalaia A, Paiva T. Sleep cycles and alpha-delta sleep in fibromyalgia syndrome. J Rheumatol. 1994 Jun;21(6):1113-7. PMID 7932424
- [Result] Drewes AM. Pain and sleep disturbances with special reference to fibromyalgia and rheumatoid arthritis. Rheumatology (Oxford). 1999 Nov;38(11):1035-8. doi: 10.1093/rheumatology/38.11.1035. No abstract available. PMID 10556252
- [Result] Flodin P, Martinsen S, Lofgren M, Bileviciute-Ljungar I, Kosek E, Fransson P. Fibromyalgia is associated with decreased connectivity between pain- and sensorimotor brain areas. Brain Connect. 2014 Oct;4(8):587-94. doi: 10.1089/brain.2014.0274. Epub 2014 Aug 7. PMID 24998297
- [Result] Napadow V, Harris RE. What has functional connectivity and chemical neuroimaging in fibromyalgia taught us about the mechanisms and management of 'centralized' pain? Arthritis Res Ther. 2014;16(5):425. doi: 10.1186/s13075-014-0425-0. PMID 25606591
- [Result] Rains JC, Penzien DB. Sleep and chronic pain: challenges to the alpha-EEG sleep pattern as a pain specific sleep anomaly. J Psychosom Res. 2003 Jan;54(1):77-83. doi: 10.1016/s0022-3999(02)00545-7. PMID 12505558
- [Result] Schmidt-Wilcke T, Ichesco E, Hampson JP, Kairys A, Peltier S, Harte S, Clauw DJ, Harris RE. Resting state connectivity correlates with drug and placebo response in fibromyalgia patients. Neuroimage Clin. 2014 Sep 16;6:252-61. doi: 10.1016/j.nicl.2014.09.007. eCollection 2014. PMID 25379438